CLINICAL TRIAL: NCT07246369
Title: The Role of Therapeutic Ultrasound in Comparison With Electrical Dry Needling in Chronic Low Back Patients Post Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/493/08/24
Record Dates: First submitted 2025-08-26; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-09

CONDITIONS: Chronic Low Back Pain (CLBP); Post Cesarean Section Patient
Keywords: Low back pain; Post cesarean section; Post partum back pain
MeSH Terms: conditions — Low Back Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Electrical Dry Needling) (Experimental)
  Interventions: Other: Electrical Dry Needling
- Group B (Therapeutic Ultrasound) (Active Comparator)
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Electrical Dry Needling — Patients in the electrical dry-needling received two 30-minute sessions per week for 6 weeks. Twenty minutes of Electrical stimulation targeted active and latent myofascial trigger points in the quadratus lumborum, multifidus, and iliocostalis muscles following MTrP. Needle insertion sites were varied based on the therapist's assessment of MTrP activity. Needles (0.25 mm × 30 mm or 0.30 mm × 40 mm) were sterilized and inserted into the trigger points, reaching the taut bands and causing local twitch responses. Needles were connected to a TENS device generating a low-frequency current (2 Hz) with a pulse duration of 250 μs and a continuous biphasic waveform, set to a "mild to moderate" intensity as reported by the patient. The 10 minutes of stretching of the quadratus lumborum, multifidus, and iliocostal muscles, including seated side stretches, cat-cow, and child's pose, improve muscle flexibility and reduce tension. (Lara-Palomo et al., 2022)
  Arms: Group A (Electrical Dry Needling)
Other: Ultrasound — In this study, participants received 12 sessions over 6 weeks, each lasting 30 minutes. The therapeutic ultrasound group received 20 minutes of continuous ultrasound using the Enraf Nonius Sonoplus 434 at 1 MHz frequency and 1.5 W/cm² intensity, applied with slow circular movements over the lower back. Treatment duration was calculated based on the area of pain using Grey's formula. Both groups also participated in a semi-supervised exercise program, starting with 10 minutes of stretching exercises for the lower back and abdominal muscles (quadratus lumborum, multifidus, and iliocostal muscles including seated side stretch, cat-cow, and child's pose improve muscle flexibility and reduce tension.) as guided by the physiotherapist. Patients were encouraged to stay active daily, perform exercises correctly, and avoid other pain treatments during the study. After completing the treatment sessions, patients continued the exercise for progress assessment until the follow-up session. (Gocevsk
  Arms: Group B (Therapeutic Ultrasound)

SUMMARY:
HYPOTHESIS

Null Hypothesis (HO):

There was a non-significant difference in the role of therapeutic ultrasound in comparison with electrical dry needling in chronic low back patients post cesarean-section.

Alternative Hypothesis (HA):

There was a significant difference in the role of therapeutic ultrasound in comparison with electrical dry needling in chronic low back patients post cesarean-section.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 25-35 years.
* History of cesarean section with epidural anesthesia
* Within the past 6 months to 8 months.
* Primiparous, postpartum women.
* Chronic low back pain persisting for more than 3 months.
* Pain intensity of at least four on a Numeric Pain Rating Scale (NPRS).

Exclusion Criteria:

* Previous low back surgery.
* Multiparous, postpartum women.
* History of Fracture (pubic fractures, vertebral fracture) and osteoporosis
* Having a stillborn fetus or lethal induction of labor.
* Severe comorbid conditions (e.g., uncontrolled diabetes, cardiovascular disease).
* Patients who experienced a C-section with general anesthesia

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline to 6 Week
  Participants in the study expressed the severity of their pain using a 10 Numeric Pain Rating Scale (NPRS). Participants are instructed to locate their level of pain on a 10-mm horizontal line, with 0 mm representing "no pain" and 10 mm representing "the most severe pain."
Tampa Scale for Kinesiophobia (TSK) | Baseline to 6 Week
  It is a measurement tool used to assess individuals' fear of movement and re-injury. This 17-item questionnaire is designed to determine an individual's fear of movement and the possibility of (re)injury. Patients evaluate their beliefs on their kinesiophobia using a 4-point scale that spans from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Al-Husban N, Elmuhtaseb MS, Al-Husban H, Nabhan M, Abuhalaweh H, Alkhatib YM, Yousef M, Aloran B, Elyyan Y, Alghazo A. Anesthesia for Cesarean Section: Retrospective Comparative Study. Int J Womens Health. 2021 Feb 2;13:141-152. doi: 10.2147/IJWH.S292434. eCollection 2021. PMID 33564269
- [Background] Al-Boloushi Z, Gomez-Trullen EM, Arian M, Fernandez D, Herrero P, Bellosta-Lopez P. Comparing two dry needling interventions for plantar heel pain: a randomised controlled trial. BMJ Open. 2020 Aug 20;10(8):e038033. doi: 10.1136/bmjopen-2020-038033. PMID 32819949
- [Background] A Abdel Hady D, Abd El-Hafeez T. Utilizing machine learning to analyze trunk movement patterns in women with postpartum low back pain. Sci Rep. 2024 Aug 12;14(1):18726. doi: 10.1038/s41598-024-68798-6. PMID 39134567